CLINICAL TRIAL: NCT04754828
Title: A Study of Bedside Versus Hallway Rounding for Neurology Inpatient Teams
Brief Title: A Study of Bedside Versus Hallway Rounding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Tracey Milligan, Neurologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2019P002584
Record Dates: First submitted 2021-02-05; First posted 2021-02-15 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Education, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bedside (Active Comparator): The bedside rounding team will perform patient presentations at the bedside, with a focus on the patient, and will ensure nursing involvement when rounding on each patient,
  Interventions: Other: Assigned to a rounding style
- Hallway (Active Comparator): The hallway rounding team will present patients outside of the patient's room, without an emphasis on nurse participation.
  Interventions: Other: Assigned to a rounding style

INTERVENTIONS:
Other: Assigned to a rounding style — Team rounded on new admissions either in hallway or at the bedside

SUMMARY:
The purpose of this study is to compare bedside rounding with hallway and conference room rounding on the neurology inpatient ward service at an academic hospital and identify best practices associated with educational and patient care outcomes. Specifically, this study will determine which rounding practices are associated with a positive educational experience for learners, greatest patient and care team communication, and time efficiency.

DETAILED DESCRIPTION:
This study will evaluate the efficacy of bedside rounding and compare it to hallway and conference room rounding on the neurology ward service at the Brigham and Women's Hospital (BWH). The neurology ward service consists of two teams, each with 10-15 vascular neurology and general neurology patients. The teams perform daily attending rounds.

Each team consists of an attending physician, a senior supervisory resident, two junior residents, several rotating residents and interns from other departments, medical students, as well as a physician assistant who alternates daily between the teams. Neurology attendings spend two weeks at a time on a team.

During a two-week attending rotation, we plan to designate one of the teams as the "bedside rounding team" and the other team as the "hallway rounding team", which will serve as the control group. The bedside rounding team will carry out patient presentations at the bedside, with a focus on the patient, while ensuring nursing involvement in each patient's room. The hallway rounding team ("the usual method") will present patients outside of the patient's room, without an added emphasis on nurse participation. Halfway through the two-week rotation, the team designation will switch in a crossover fashion, so that the initial bedside rounding team will become the hallway rounding team, and vice versa. Our planned study period is Monday through Friday for a consecutive 6-8 week period, and we anticipate including about 150-200 patients in our study.

To evaluate staff educational experience, patient and interprofessional communication, and clinical care outcomes of these two rounding approaches, we plan to survey patients, resident trainees, attendings, and nurses on both teams. For collection of data, a student observer or research assistant familiar with the study purpose and methods will accompany a neurology team during weekday morning rounds and record data about the composition and timing of rounds.

Eligible participants include adult patients and providers (nurses; physicians, including residents and attendings; and ancillary providers) involved in the inpatient neurology service at BWH. Patients whose primary language is English will be included in the study with notation of this feature. Observations will focus on activities of the physician providers. Surveys for medical education will involve physician participants who give consent. Surveys of patient care and communication will involve patients and nurses who give consent.

ELIGIBILITY:
Inclusion Criteria:

* new admission to neurology team

Exclusion Criteria:

* comfort measures as sole treatment goal

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Mean patient rounding time as assessed by time-motion analysis | 90 days
  The first primary outcome measure will be mean rounding time in minutes per patient in the bedside and hallway groups.
Mean rounding proportion spent at the patient's bedside as assessed by time-motion analysis | 90 days
  The second primary outcome measure will be mean rounding proportion in percent spent at the patient's bedside in the bedside and hallway groups
Mean rounding proportion spent on various rounding activities as assessed by time-motion analysis | 90 days
  The third primary outcome measure will be mean rounding proportion in percent spent on history taking, review of data such as imaging, physical exam, answering patient questions, teaching, and discussion of plan in the bedside and hallway groups

SECONDARY OUTCOMES:
Patient, nurse, resident, and attending physician satisfaction with rounds as assessed by surveys | 90 days
  The secondary outcome will be patient, nurse, resident, and attending physician satisfaction with and perception of rounds as assessed by surveys using a 5-point Likert scale with 5 being the highest satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham Health, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Solomon JM, Bhattacharyya S, Ali AS, Cleary L, Dibari S, Boxer R, Healy BC, Milligan TA. Randomized Study of Bedside vs Hallway Rounding: Neurology Rounding Study. Neurology. 2021 Aug 31;97(9):434-442. doi: 10.1212/WNL.0000000000012407. Epub 2021 Jun 22. PMID 34158383